CLINICAL TRIAL: NCT04494789
Title: A Phase II Open Label Randomised Controlled Clinical Trial of Different Dosing Regimens of Fludrocortisone in Septic Shock With Assessment of Temporal Changes in Hormonal, Inflammatory, and Genetic Markers of Vascular Responsiveness
Brief Title: Fludrocortisone Dose Response Relationship in Septic Shock - FluDReSS
Acronym: FluDReSS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The George Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GI-CC35837377
Record Dates: First submitted 2020-07-19; First posted 2020-07-31 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Critically Ill; Septic Shock
MeSH Terms: conditions — Critical Illness; Shock, Septic | interventions — fludrocortisone acetate; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Fludrocortisone dosing regime: 24hrs (Active Comparator): Receive 50mcg doses of fludrocortisone every 24hrs
  Interventions: Drug: Fludrocortisone Acetate
- Fludrocortisone dosing regime: 12hrs (Active Comparator): Receive 50mcg doses of fludrocortisone every 12hrs
  Interventions: Drug: Fludrocortisone Acetate
- Fludrocortisone dosing regime: 6hrs (Active Comparator): Receive 50mcg doses of fludrocortisone every 6hrs
  Interventions: Drug: Fludrocortisone Acetate
- Control Arm (Placebo Comparator): Receives standard treatment without fludrocortisone dosing regime
  Interventions: Other: Standard Therapy

INTERVENTIONS:
Drug: Fludrocortisone Acetate — 50mcg
  Arms: Fludrocortisone dosing regime: 24hrs
Drug: Fludrocortisone Acetate — 100mcg
  Arms: Fludrocortisone dosing regime: 12hrs
Drug: Fludrocortisone Acetate — 200mcg
  Arms: Fludrocortisone dosing regime: 6hrs
Other: Standard Therapy — NO Fludrocortisone
  Arms: Control Arm

SUMMARY:
The purpose of this study is to determine the most suitable dose of Fludrocortisone in reversal of sepsis and shock associated with sepsis in patients who are admitted to the ICU.

The investigators will be looking to see whether patients receiving Fludrocortisone at different doses recover quicker and spend less time in hospital and in ICU, and to understand the reasons why this happens at certain doses.

Sepsis is caused by toxic substances (toxins) from bacteria and other organism entering the bloodstream from a site of infection. In some people, the infection can progress to sepsis and septic shock where the functions of organs in the body are affected. Patients suffering from sepsis and septic shock are commonly managed in the intensive care unit (ICU) where they are prescribed antibiotics as standard therapy, as well as other therapies to support the functions of the body.

Fludrocortisone is a steroid that has previously shown to be beneficial to help in shock in patients in ICU, but more information is required about the exact dose that is required to achieve this. This has been shown by previous research.

However, the exact role of Fludrocortisone and the best dose has not been studied adequately to date as well as the ways in how it works within the body. The study aims to look tat the dose and the way it works.

DETAILED DESCRIPTION:
Aim:

1. To conduct a multi-centre randomised controlled trial to assess the effect of 3 different dose regimens of fludrocortisone on shock reversal in septic shock patients treated with hydrocortisone.
2. To assess the temporal changes in endocrine inflammatory and gene expression markers in septic shock patients.

Hypotheses:

In patients with septic shock treated with hydrocortisone,

1. The addition of fludrocortisone to hydrocortisone results in improved vascular responsiveness to vasopressors as compared to hydrocortisone alone
2. The improvement of vascular responsiveness with fludrocortisone is in a dose dependent manner
3. Enterally administered fludrocortisone results in adequate plasma level
4. Patients who have early reversal of shock have higher concentrations of, angiotensin II and angiotensin II-receptor expression and reduced angiotensin converting enzyme 2 (ACE 2) concentrations at baseline and throughout the course of their illness
5. Patients who have early reversal of shock have higher concentrations of plasma free cortisol, aldosterone and glucocorticoid and mineralocorticoid receptor expression at baseline and throughout the course of their illness.
6. Patients who demonstrate evidence of both greater angiotensin II and glucocorticoid receptor expression will have earlier shock reversal than those who have an increase in expression of either of these receptors.
7. There is a different temporal change in the plasma concentrations and receptor expression profiles in early shock reversal patients vs. delayed shock reversal patients.

   300 patients will be recruited and randomised to enteral doses of 50mcg fludrocortisone Q24H, Q12H, Q6H or to the control arm of the study. The study will enrol patients admitted to a participating intensive care unit and who meet all the inclusion criteria and no exclusion criteria. Patients in a fludrocortisone arm will receive enteral fludrocortisone for a maximum of 7 days or until sustained shock reversal or until discharge from ICU whichever is earlier.

   Blood samples acquired will be analysed for:
   * Endocrine - Cortisol, free cortisol, aldosterone and metabolites
   * Inflammatory - Cytokine profiles, markers of vasoplegia
   * Gene Expression - Whole genome RNA sequencing and single cell sequencing
   * To assess the plasma levels following enteral administration of fludrocortisone in all patients enrolled to undertake detailed analysis of fludrocortisone kinetics in a subgroup of 30 patients enrolled (10 patients in each dosing group).

   For all patients, data will be collected at baseline and daily whilst in the ICU for up to 8 days. Patients will be followed up to time of discharge from hospital or day 28 if they are still in hospital, whichever occurs first

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older
2. Documented site, or strong suspicion of infection with 2 of the 4 clinical signs of inflammation:

   1. Core temperature > 38oC or < 35oC
   2. Heart rate > 90bpm
   3. Respiratory rate > 20bpm, or PaCO2 < 32mmHg, or mechanical ventilation
   4. White cell count > 12 x 109/L or < 4 x 109/L or > 10% immature neutrophils\
3. Being treated with Hydrocortisone at a daily dose of 200mg / day as adjunctive treatment for sepsis
4. Being treated with mechanical ventilation at the time of randomisation (includes mask BiPAP/CPAP)
5. Being treated with continuous vasopressors or inotropes to maintain a systolic blood pressure > 90mmHg, or mean arterial pressure > 60mmHg or a MAP target set by the treating clinician for maintaining perfusion
6. Administration of vasopressors or inotropes for > 4 hours and present at time of randomisation

Exclusion Criteria:

1. Met all inclusion criteria more than 24 hours ago
2. Patients taking long term corticosteroids or fludrocortisone
3. Patients with systemic fungal infection
4. Death is deemed inevitable or imminent during this admission and either the attending physician, patient or surrogate legal decision maker is not committed to active treatment
5. Patient unable to receive enteral medication
6. Death from underlying disease likely within 90 days
7. Patient has been previously enrolled in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2021-02-11 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Time to resolution of shock by Intervention group allocation | 7 DAYS
  To the assess the time it takes for shock to resolve in each intervention arm
Time to resolution of shock and Fludrocortisone Levels | 7 days
  Assess the levels of fludrocortisone in the interventional groups at time of resolution of shock
Vasopressor Responsiveness by Intervention group allocation | 7 days
  Area under the curve of vasopressor dose in each intervention arm
Vasopressor Responsiveness and Fludrocortisone Levels | 7 days
  Area under the curve of vasopressor dose associated with fludrocortisone levels

SECONDARY OUTCOMES:
Recurrence of shock | censored at day 28
  Time between a new episode of shock after reversal of the initial episode
Ventilation free days | censored at day 28
  Number of Days that are without ventilation during admission
ICU and hospital length of Stay | censored at day 28
  Total number of days in ICU and in hospital for the index admission
ICU and hospital mortality | censored at day 28
  The number of deaths that are recorded in participants and the location of the deaths when in hospital - ICU or ward. This will include cause of death
Delta SOFA Score | censored at day 28
  Baseline SOFA score to SOFAmax - numerical calculation based on scoring system of each participant during their admission
Maximal SOFA score | censored at day 28
  Maximum SOFA score for each participant during their admission
Superinfection | censored at day 28
  This is the number of new infections that occur >48hrs after commencing study drug

OTHER OUTCOMES:
Pharmacokinetic Outcome To assess the plasma levels of enterally administered fludrocortisone in all patients enrolled | 7 days
  Time to peak concentration of Fludrocortisone
Pharmacokinetic Outcomes - To undertake detailed analysis of fludrocortisone kinetics in a subgroup of 30 patients enrolled (10 patients in each dosing group) | 7 days
  Time to absorption, clearance and metabolism of fludrocortisone in participants in each intervention arm except for the control arm
Vascular Responsiveness Analysis | 7 days
  Acquisition of blood samples at 4 timepoints over the first 7 days or until discharge from ICU for exploratory analysis to assess a range of biomarkers and their interactions with the primary outcomes

CONTACTS AND LOCATIONS:
Overall Officials: James Walsham, MB ChB, MRCP, FCICM., Principal Investigator — Princess Alexandra Hospital
Locations (9):
- Australia (9):
  - Blacktown Hospital, Sydney, New South Wales
  - Royal North Shore Hospital, Sydney, New South Wales
  - Royal Brisbane Women's Hospital, Brisbane, Queensland
  - Wesley Hospital, Brisbane, Queensland
  - Gold Coast University Hospital, Gold Coast, Queensland
  - Mater Misericordiae, Raymond Terrace, Queensland
  - Princess Alexandra Hospiital, Woolloongabba, Queensland
  - Queen Elizabeth II Hospital, Adelaide, South Australia
  - Austin Hospital, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: Undecided